CLINICAL TRIAL: NCT03601884
Title: Effectiveness of Optimal Health Program in Improving Self-efficacy in Patients With Diabetes Mellitus in Putrajaya, Malaysia
Brief Title: Effectiveness of OHP in Improving Self-efficacy in Patients With Diabetes Mellitus
Acronym: OHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Aida Farhana Suhaimi, Clinical Psychologist, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHPMALAYSIA
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus; Chronic Illness
Keywords: Well-being; Self-efficacy; Self-management; Psychosocial; Malaysia
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is a Randomised Controlled Trial. The sampling frame will be patients with diabetes registered in all the government health clinics located in Putrajaya. Patients are screened at the beginning and later interviewed using a structured questionnaire and intake interview. All four Health Clinics in Putrajaya will participate in the study, randomization will be conducted at the facility level.
  This study is a two arm - experimental vs. control group RCT. Participants are randomly allocated at facility level. All four health clinics will be randomly assigned to the OHP and TAU (experimental group) or TAU (control group), with two health clinics randomly allocated in the experimental group and another two the control group.
Who Masked: Participant
Masking Description: To reduce performance bias after the randomization process, blinding is adopted. However, due to the conflicting requirements of ethical and methodological aspects in designing a randomized controlled trial with a psychosocial intervention, double blinding and randomizing each individual participant posits a huge challenge. Patients, the attending doctors and the co-author involved in randomly assigning the group will be blinded in a way that none of them will know which group is considered the experimental group and the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OHP and Treatment as usual (TAU) (Experimental): Optimal Health Program (OHP) A self-management program that promotes patients to be actively involved in their own healthcare and overall well-being through enhancing self-efficacy.
  Treatment is delivered by a trained facilitator in OHP. The OHP is delivered in groups of 8 to 10 participants It consists of 5 weekly, 1.5 hour sessions and an additional booster session post-program at 3 months a The group facilitator will contact the participants by phone at 8 weeks and 16 weeks.
  Treatment-as-usual TAU is the pharmacological treatment received or prescribed by the patients' attending doctor.
  To ensure standardization of treatment, attending doctors will be reminded to manage patients in accordance with the Clinical practice Guideline in Managing Diabetes Melllitus in adult patients.
  Interventions: Behavioral: Optimal Health Program; Other: Treatment as Usual
- TAU Alone (Other): Treatment-as-usual TAU is the pharmacological treatment received or prescribed by the patients' attending doctor.
  To ensure standardization of treatment, attending doctors will be reminded to manage patients in accordance with the Clinical practice Guideline in Managing Diabetes Melllitus in adult patients.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Optimal Health Program — The Optimal Health Program (OHP) is a self-management psychosocial program that promotes patients to be actively involved in their own healthcare and overall well-being. Sessions include Optimal Health, I-CAN-DO Model, Medication & Metabolic Monitoring, Collaborative & Strategies, Change enhancement, Visioning & Goal Setting and Maintain Well-being.
  Other Names: OHP; Wellbeing Psychosocial Program
  Arms: OHP and Treatment as usual (TAU)
Other: Treatment as Usual — Treatment-as-usual TAU is the pharmacological treatment received or prescribed by the patients' attending doctor.
  To ensure standardization of treatment, attending doctors will be reminded to manage patients in accordance with the Clinical practice Guideline in Managing Diabetes Melllitus in adult patients.
  Other Names: TAU

SUMMARY:
Addressing the increasing trend in diabetes and mental illness co-morbidities, Malaysia is currently in need of a self- management program that promotes patient empowerment and overall well-being - beyond education. Committing to the self-care behaviours is highly dependent on the individual's self-efficacy. Self-efficacy has been shown to have a direct positive relationship with self-care behaviours, direct negative relationship with psychological distress and depression. Self-efficacy has also been found to hold a mediating effect on the relationship between emotional distress and self-care behaviours.

The objective of this study is to assess the effectiveness of a self-management program for patients with diabetes, the Optimal Health Program (OHP) in improving self-efficacy, depression, anxiety, diabetes distress, well-being and self-care. This study is a randomized controlled trial study of patients with diabetes attending the four diabetes health clinics within the Putrajaya District. Eligible patients will be randomly allocated to either treatment as usual (TAU) or OHP and treatment as usual (OHP + TAU). The treatment as usual group (TAU) participants will be invited to participate in the OHP at the end of the study. The participants in the OHP + TAU will attend 5 weekly 1.5 hour sessions and a booster session at 3 months. Following ethics approval, recruitment and training will commence in September, data collection expected to be until April 2020.

It is hypothesized that the OHP + TAU group will have higher self-efficacy, well-being and self-care scores and reduced depression, anxiety, diabetes related-distress and HbA1c. This study will contribute towards the gap in the literature in the effectiveness of a self-efficacy enhancing psychosocial self-management program among diabetes patients in Malaysia within a primary care setting.

DETAILED DESCRIPTION:
Background and Significance

Diabetes currently affects 1 in 5 adults, with the most affected within the productive age span and an expectation of continual increase in the future. Mirroring the global trend, Malaysia has approximately 2.6 million adults having diabetes mellitus in Malaysia with an up to 31% increase from 2006 to 2011. The complexity of diabetes mellitus itself is associated with not just the physical health but also the patients' emotional well-being and mental health, social, occupational and overall quality of life. The current blooming diabetes population with increasing psychosocial barriers brings about a huge impact on the complexity of diabetes. Psychosocial self-management is central to effective management in diabetes. Nonetheless, committing to the self-care behaviours is highly dependent on the individual's self-efficacy.

Self-efficacy is the individual's belief about their capabilities to cope and manage their diabetes. Self-efficacy can be assessed based on the individual's perceived ability - (1) to conduct the specific diabetes self-care activities and (2) to manage their psychosocial issues related to diabetes psychosocial self-efficacy. Self-efficacy has been shown to have a direct positive relationship with self-care behaviours 4, direct negative relationship with psychological distress and depression. Self-efficacy has also been found to hold a mediating effect on the relationship between emotional distress and self-care behaviours.

Addressing the increasing trend in diabetes and mental illness comorbidities, Malaysia is currently in need of a self- management program that promotes patient empowerment and overall well-being - beyond education. With limited mental health professionals and resources, there is a greater need to build the capacity of the health care system especially within the primary care setting. A low intensity intervention program that plays a preventative as well as a curative role conducted within the primary care setting would be of great significant.

Based on the theory of Self-Efficacy, the Optimal Health Program (OHP) is a self-efficacy enhancing management program that promotes patients to be actively involved in their own healthcare and overall well-being. The aim of OHP is to improve a person's health literacy and overall wellbeing through self-efficacy and understanding their strengths and vulnerabilities. Evidently, OHP has shown to be effective in improving health and social functioning in mental health patients, substance use and psychotic disorders. The OHP has slowly expanded towards managing physical health and chronic illnesses. Due to its holistic approach by addressing multiple areas of an individual's life creates tremendous potential in the management of the complexity of chronic illness.

OHP will be the first engagement tool in Malaysia that will allow health care professionals to address the mental health issues and promote overall wellbeing in these chronic ill patients. OHP is a low intensity intervention program that can be delivered by trained facilitators. The delivery of self-management programs has been shown to be equally effective when delivered by diabetes educators, peers, practice staffs as well as specifically trained program facilitators.

Through the OHP it is hope that it will provide a low intensity intervention program for early intervention within the primary care setting that can be delivered by a broad range of health care providers. It offers a platform for wide range of health care providers within the primary care to engage in a discussion with patients regarding their well-being through a patient centered collaborative approach.

Additionally, in 2015, the 5th edition CPG Management of Diabetes Mellitus Type 2 was issued. The standard of practice especially within the primary health care is greatly guided by the National Clinical Practice Guideline (CPG). The latest CPG puts a greater emphasis in early screening and detection inclusive of mental health issues and patient centered care. With this greater emphasis, it is worthwhile to further examine the effectiveness of the current standard of practice as guided by the latest version of the CPG or whether an add-on psychosocial self-management program to the current practice would yield greater impact.

Significance of study

Based on the National Health Morbidity Survey 2015, the prevalence for diabetes in Putrajaya was reported to be above the national prevalence and at the top half highest prevalence for diabetes (19.2%) as compared to all the states in Malaysia, Moreover, Putrajaya had the highest prevalence for overweight (37%) and abdominal obesity, obesity I, obesity II as well as obesity III (25.8%). Despite that, Putrajaya was found to have the second highest prevalence for adequate health literacy (16%).

Even though the understanding and knowledge on ways to promote and maintain good health was comparably high, prevalence of diabetes and obesity were still at large. This may imply a dissonance between being educated on the illness and the ability to utilize the knowledge to commit to healthy lifestyle changes. Enhancing self-efficacy links this dissonance - that is by improving people's beliefs of their own capabilities to self-manage their diabetes and to produce an impact in their lives.

Therefore, this study will contribute towards the gap in the literature in the effectiveness of a self-efficacy enhancing psychosocial self-management program among diabetes patients in Malaysia. The OHP provides an engagement tool that works as a curative and preventative role for primary health care providers. The OHP is a low-intensity, structured, psychosocial program that emphasizes well-being as compared to illness that is suitable to be given within a primary health care setting .

Specifically, it will be looking at the effectiveness of OHP and treatment-as-usual (TAU) as compared to TAU alone, in improving self-efficacy in patients with diabetes that are currently attending the health clinics within the Putrajaya district. In addition, it will also examine the effectiveness of OHP in improving anxiety, depression, diabetes-related distress, self-care behaviours and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* patients with a known diagnosis of Diabetes Mellitus Type 2 given by their attending physicians,
* aged between 18 to 65 years old
* currently attending the health clinics in Putrajaya.
* able to provide consent independently without assistance.

Exclusion Criteria:

* patients that are not able to write and read,
* does not understand Malay or English,
* has a serious acute medical illness (e.g. delusional, delirium) during the intake.
* Patients who are currently attending intensive psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in Diabetes Empowerment Scale (DES) scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  Diabetes Empowerment Scale (DES) An 8 item self-administered measurement that assesses the overall diabetes-related psychosocial self-efficacy. All 8 items are rated from 0 (strongly disagree) to 4 (strongly agree). The sum of all items ranged from 0 to 32. Higher scores indicate greater psychosocial self-efficacy.
Difference in Diabetes Management Self-Efficacy Scale (DMSES) scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  A 20-item self-administered measurement that assess self-efficacy in managing specific diabetes self-care behaviours. All items are rated between 0 (Not at all confident) to 10 (totally confident).
  The sum of all items range between 0 (no self-efficacy) to 100 (very high self-efficacy).

SECONDARY OUTCOMES:
Difference in PHQ scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  9 item self-administered measurement that assess depression
Difference in GAD scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  7 item self-administered measurement that assess depression
Difference in PAID-20 scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  20 item self-administered measurement that assess diabetes related distress.
Difference in WHO-5 scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  5 item self-administered measurement that assess wellbeing
Difference in diabetes self-care behaviours scores between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 5, Week 18, Week 30
  10 item self-administered measurement that assess diabetes self-care behaviours
Difference in HbA1c between OHP+TAU (experimental group) and TAU alone (control group), and within OHP plus TAU across time | Week 1, Week 30
  Glycaemic control as assessed by HbA1c level

CONTACTS AND LOCATIONS:
Overall Officials: Aida F Suhaimi, Ms, Principal Investigator — Universiti Putra Malaysia
Locations (4):
- Malaysia (4):
  - Klinik Kesihatan Presint 11, Putrajaya
  - Klinik Kesihatan Presint 14, Putrajaya
  - Klinik Kesihatan Presint 18, Putrajaya
  - Klinik Kesihatan Presint 9, Putrajaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suhaimi AF, Ibrahim N, Tan KA, Silim UA, Moore G, Ryan B, Castle DJ. Effectiveness of a culturally adapted biopsychosocial intervention (POHON SIHAT) in improving self-efficacy in patients with diabetes attending primary healthcare clinics in Putrajaya, Malaysia: study protocol of a randomised controlled trial. BMJ Open. 2020 Feb 16;10(2):e033920. doi: 10.1136/bmjopen-2019-033920. PMID 32066607